CLINICAL TRIAL: NCT02556086
Title: A Phase 2b Evaluation of Daclatasvir/Sofosbuvir in Non-Cirrhotic Treatment Naive Subjects With Genotype 1, 2, 3 and 4 Chronic Hepatitis C Virus Coinfected With Human Immunodeficiency Virus (HIV-1)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AI444-378; 2015-003467-12 (EudraCT Number)
Record Dates: First submitted 2015-09-15; First posted 2015-09-22 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2015-11

CONDITIONS: Hepatitis C
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; Sofosbuvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Daclatasvir + Sofosbuvir (Experimental): Daclatasvir 30, 60, 90 mg tablet (dose is dependent on cART regimen) + Sofosbuvir 400 mg tablet oral dosing once daily for 8 weeks
  Interventions: Drug: Daclatasvir; Drug: Sofosbuvir

INTERVENTIONS:
Drug: Daclatasvir
Drug: Sofosbuvir

SUMMARY:
The purpose of the study is to determine if combination therapy with daclatasvir (DCV) and sofosbuvir (SOF) for 8 weeks is safe and effective in patients who have never been treated previously without liver cirrhosis who are chronically infected with hepatitis C virus (HCV)/HIV-1 Coinfection genotype (GT) 1, 2, 3, 4 patients.

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* HCV RNA < 2000000 IU/mL
* Never taken medication for HCV
* No Liver Cirrhosis
* No advanced fibrosis
* Body mass index(BMI) 18-40 kg/m^2
* Genotype 1-4

Exclusion Criteria:

* Infection with HCV other than GT-1, 2, 3 or GT-4 or subjects with mixed infections of any genotype
* Evidence of decompensated liver
* Subjects Infected with HIV 2
* Hepatitis B virus (HBV) coinfection
* Liver Cirrhosis
* Advanced fibrosis (F3-F4)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with SVR12 | Post treatment follow-up week 12
  SVR12 rate defined as HCV RNA < LLOQ target detected (TD) or target not detected (TND) at follow-up Week 12 in subjects infected with HCV/HIV-1 coinfection genotype 1-4

SECONDARY OUTCOMES:
Sustained virologic response (SVR12) rate | Approximately 2 years
  SVR12 rate defined as HCV RNA < lower limit of quantification (LLOQ) target detected (TD) or target not detected (TND) at follow-up Week 12 in subjects infected with HCV/HIV-1 coinfection, by individual genotype (1-4)
Treatment safety measured by the number of incidence of serious adverse event (SAEs), discontinuations due to adverse event (AEs), Grade 3/4 AEs and Grade 3/4 clinical laboratory abnormalities through the end of treatment | Approximately 2 years
Proportion of subjects who achieve HCV RNA < LLOQ-TD/TND at each of the following Weeks: 1, 2, 4, 6, 8, EOT, post-treatment Week 4 in subjects on the 8-week regimen of DCV/SOF | Approximately 2 years
Proportion of subjects who achieve HCV RNA < LLOQ TND at each of the following Weeks: 1, 2, 4, 6, 8, end of treatment (EOT), in subjects on the 8-week regimen of DCV/SOF | Approximately 2 years
Proportion of subjects receiving cART who maintain HIV virologic suppression | Approximately 2 years
Proportion of subjects receiving cART who experience HIV virologic failure | Approximately 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (13):
- Canada (8):
  - Local Institution, Edmonton, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Victoria, British Columbia
  - Local Institution, Ottawa, Ontario
  - Local Institution, Toronto, Ontario
  - Local Institution, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution, Regina, Saskatchewan
- France (5):
  - Local Institution, Marseille
  - Local Institution, Nantes
  - Local Institution, Nice
  - Local Institution, Paris
  - Local Institution, Pessac

REFERENCES:
- See also: BMS clinical trial educational resource — http://www.bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx